CLINICAL TRIAL: NCT00190567
Title: Biomechanical Effects of Duloxetine on Bladder Function and Sphincter Resistance During the Emptying Phase and on Urethral Function During the Filling Phase of the Micturition Cycle in Women With Pure Genuine Stress Incontinence
Brief Title: Biomechanical Effects of Duloxetine on Bladder and Sphincter Muscle Function in Women in Pure Genuine Stress Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2595; F1J-MC-SBAB
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Urinary Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine
Drug: Placebo

SUMMARY:
Double-blind placebo-controlled study of the biomechanical effects of duloxetine compared with placebo in the treatment of women with pure genuine stress incontinence

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between 18 and 75 years of age
* Diagnosis of GSI
* Have discrete episodes of incontinence

Exclusion Criteria:

* Positive urine culture at visit 1
* Use of MAOI
* Have had continence or urethral surgery
* Use of anti-incontinence device, vaginal pessaries or medications for the treatment of urinary incontinence
* Began pelvic floor muscle exercises within 6 months prior to study entry.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2001-10; Study Completion 2006-04

PRIMARY OUTCOMES:
Compare the effects of duloxetine with placebo in women with urodynamically proved genuine stress incontinence(GSI)on vesical Valsalva leak point pressure

SECONDARY OUTCOMES:
Compare the effects of duloxetine with that of placebo on measures of bladder emptying phase function derived from
non-instrumented and instrumented uroflowmetry studies
Percent change in Incontinent Episode Frequency (IEF) from baseline to endpoint
Subject-perceived improvement in their GSI as measured by the Patient Global Impressions-Improvement (PGI-I) questionnaire at endpoint
Compare duloxetine responders with duloxetine non-responders with respect to:
Baseline measures of urethral function
Outcome measures of urethral function
Outcome measures of emptying function
Vital signs, laboratory values and the occurrence of treatment-emergent adverse events
In the open-label extension:
Determine the effects of duloxetine six to seven months after initiation on measures of urethral function
Collect long-term data on the maintenance of effect of duloxetine in the treatment of GSI as measured by IEF, PGI-I, vital signs, laboratory values and the occurrence of treatment-emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon -Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5hours, EST), or speak with your personal physician, Indianapolis, Indiana, United States